CLINICAL TRIAL: NCT07204821
Title: Functional Inspiratory Versus Expiratory Muscle Electrical Stimulation on Weaning Outcomes in Mechanically Ventilated Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayah Japer Muhammad Muhammad Abu-Bakr, physiotherapist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Icu
Keywords: Functional Inspiratory Muscle Electrical Stimulation, Functional Expiratory Muscle Electrical Stimulation, Weaning Outcomes in Mechanically Ventilated Patients.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): Inspiratory muscle FES by Flexistem Digital electrical muscle stimulator +Early rehabilitation program. The current is pulsed, biphasic, and symmetric, with Frequency of 30 hertz , Phase width of 200µs, ON time 2s: OFF time 3s. Patients will be instructed to keep their RR constant and to coordinate their breathing with the pulsing of the electrical current . Four silicone-carbon electrodes (4x4cm) were placed on the clean skin with gel. Two electrodes each will be placed above and below the right and left sides of the xiphoid process within the seventh and eighth anterior intercostal space. In addition, two electrodes each were placed on the right and left midaxillary line of the seventh and eighth anterior space Two sessions daily, each session will last for 30 minutes; the patients remained in the semi-Fowler position 30 º with the lower extremities extended and arms alongside the body
  Interventions: Device: Inspiratory muscle functional electrical stimulation by Flexistem Digital electrical muscle stimulator; Device: Early rehabilitation program
- Group B (Active Comparator): Expiratory muscle FES by Flexistem Digital electrical muscle stimulator+Early rehabilitation program. FES is applied for 30 min, two sessions daily, until patients are weaned from mechanical ventilation, but no longer than six weeks. Stimulation will be applied during exhalation and via surface electrodes on the abdominal wall Four pairs silicone-carbon electrodes (4x9cm) were placed on the clean skin with gel, and stimulation intensity will be titrated in order to activate the external oblique, internal oblique, transversus abdominis and Rectus abdominis muscles. settings are as follows: Frequency 30 Hz, pulse width 352 µs and a current intensity set to cause strong muscle contraction, with a maximum intensity initially set at 60 mA . Then we amend the protocol to allow a maximum intensity of 100 mA . Strong muscle contraction will verify (visible and palpable) every ten minutes throughout each FES session, and if necessary, stimulation intensity was increased.
  Interventions: Device: Expiratory muscle functional electrical stimulation by Flexistem Digital electrical muscle stimulator; Device: Early rehabilitation program
- Group C (Active Comparator): Inspiratory muscle functional electrical stimulation and Expiratory muscle functional electrical stimulation along with Early rehabilitation program plus medical treatment.
  Interventions: Device: Inspiratory muscle functional electrical stimulation by Flexistem Digital electrical muscle stimulator; Device: Expiratory muscle functional electrical stimulation by Flexistem Digital electrical muscle stimulator; Device: Early rehabilitation program
- Group D (Control Group) (Active Comparator): early rehabilitation program plus medical treatment
  Rehabilitation therapy which consisted of six levels:
  Level 0 turning over once every 2 h for unconscious patients with unstable vital signs level 1-2 in addition to turning over, maintaining joint range of motion to prevent muscle atrophy, and placing normal limb position for conscious patients who could sit up for at least 20 min, 2 times a day Level 3 similar to level 2, but sitting on the edge of the bed for patients who could perform upper-limb anti-gravity training Level 4 similar to level 3, but standing up or sitting in a chair for at least 20 min a day for patients who could perform lower-limb anti-gravity training Level 5 patients actively moved from the bed and walked bedside
  Interventions: Device: Early rehabilitation program

INTERVENTIONS:
Device: Inspiratory muscle functional electrical stimulation by Flexistem Digital electrical muscle stimulator — The electrical current is pulsed, biphasic, and symmetric, with the Frequency of 30 hertz, Phase width of 200µs, ON time 2s: OFF time 3s. Patients will be instructed to keep their RR constant and to coordinate their breathing with the pulsing of the electrical current. The intensity of the current is the minimum necessary to obtain diaphragm muscle contraction . Four silicone-carbon electrodes (4x4cm) were placed on the clean skin with gel. 2 electrodes each will be placed above and below the right and left sides of the xiphoid process within the seventh and eighth anterior intercostal space. In addition, two electrodes each were placed on the right and left midaxillary line of the seventh and eighth anterior intercostal space Two sessions daily, each session will last for 30 minutes; the patients remained in the semi-Fowler position 30 º with the lower extremities extended and arms alongside the body
  Arms: Group A; Group C
Device: Expiratory muscle functional electrical stimulation by Flexistem Digital electrical muscle stimulator — FES is applied for 30 min, 2 sessions daily, until patients are weaned from mechanical ventilation, but no longer than 6 weeks.Stimulation will be applied via surface electrodes on the abdominal wall Four pairs silicone-carbon electrodes (4x9cm) were placed on the clean skin with gel, and stimulation intensity will be titrated in order to activate the external oblique, internal oblique, transversus abdominis and Rectus abdominis muscles. The patient's tolerance of expiratory muscle FES is continuously monitored;Frequency 30 Hz, pulse width 352 µs and intensity set to cause strong muscle contraction, with a maximum intensity initially set at 60 mA (tolerated intensity in healthy volunteers). Then we amend the protocol to allow a maximum intensity of 100 mA .Strong muscle contraction will verify (visible and palpable) every ten minutes throughout each FES session, and if necessary, stimulation intensity was increased.
  Arms: Group B; Group C
Device: Early rehabilitation program — Rehabilitation therapy which consisted of six levels:
  Level 0 turning over once every 2 h for unconscious patients with unstable vital signs level 1-2 in addition to turning over, maintaining joint range of motion to prevent muscle atrophy, and placing normal limb position for conscious patients who could sit up for at least 20 min, 2 times a day Level 3 similar to level 2, but sitting on the edge of the bed for patients who could perform upper-limb anti-gravity training Level 4 similar to level 3, but standing up or sitting in a chair for at least 20 min a day for patients who could perform lower-limb anti-gravity training Level 5 patients actively moved from the bed and walked bedside

SUMMARY:
The Goal of This Clinical Trail is

* To find out the difference in the effect of inspiratory muscle functional electrical stimulation and expiratory muscle functional electrical stimulation on weaning outcomes mechanically ventilated patients.
* To investigate the effect of inspiratory muscle functional electrical stimulation and expiratory muscle functional electrical stimulation on Laboratory investigation (Arterial Blood Gases).
* To investigate the effect of inspiratory muscle functional electrical stimulation and expiratory muscle functional electrical stimulation on Sonar parameters (Diaphragmatic excursion, Diaphragmatic muscle fractional thickness in the end of inspiration and the end of expiration and abdominal muscles wall thickness). To evaluate the effect of inspiratory muscle functional electrical stimulation and expiratory muscle functional electrical stimulation on (ICU length of stay and Spontaneous Breathing Trail (SBT)).

DETAILED DESCRIPTION:
Type of Study: This study will be randomized clinical trial. Study Procedures: 100 mechanically ventilated both sexes patients will be recruited in this study from intensive care unit, Beni-Suef University Hospital, their ages range from 45 to 65 years.

The selected patients will be all mechanically ventilated due to respiratory failure and randomly Participants will be randomly assigned to the three study groups and one control group . We will prepare (100) identical envelops, (25) of them will be filled with a label identifying Group (A) with all instruction details, while the second (25) will be filled with a label identifying the Group (B), the third (25) will be filled with a label identifying the Group (C), the last (25) will be filled with a label identifying the Group (D). All envelops will be prepared by the investigator and sealed before starting enrollment:

1. Study group (A) include mechanically ventilated patients will receive Inspiratory muscle functional electrical stimulation along with Early rehabilitation program plus medical treatment.
2. Study group (B) include mechanically ventilated patients will receive Expiratory muscle functional electrical stimulation along with Early rehabilitation program plus medical treatment.
3. Study group (C) include mechanically ventilated patients will receive Inspiratory muscle functional electrical stimulation and Expiratory muscle functional electrical stimulation along with Early rehabilitation program plus medical treatment.
4. Control group (D) include mechanically ventilated patients will receive early rehabilitation program plus medical treatment.

A) Measurement procedures:

1. ICU length of stay: The number of days from ICU admission to ICU discharges
2. Monitoring :

   * Mode of ventilation parameters:

     i) Fiao2 ii) PEEP iii) Tidal Volume iv) Respiratory Rate v) Maximum Respiratory Pressure
   * The Duration and Type of Weaning:

   The Classification of patients according to the weaning process: Classification of patients according to the difficulty and length of the weaning process into 3 Groups: 1- Simple weaning Patients who proceed from initiation of weaning to successful extubation on the first attempt without difficulty 2- Difficult weaning Patients who fail initial weaning and require up to three SBT or as long as 7 days from the first SBT to achieve successful weaning 3- Prolonged weaning Patients who fail at least three weaning attempts or require 7 days of weaning after the first SBT
3. Laboratory investigation :

   Arterial Blood Gases (ABG): ABG may show hypoxemia that increased oxygen supplementation and hypercapnia. The analysis will be used as initial evaluation 10 minutes before the session and final evaluation 20 minutes after the end of the session. The samples will be drawn from radial artery with a preheparinized syringe. All the samples will be analyzed for: pH, PaO2, SaO2, PaCO2, and HCO3.
4. Sonar parameters:

   * Diaphragmatic excursion.
   * Diaphragmatic muscle fractional thickness in the end of inspiration and the end of expiration.
   * Abdominal muscles wall thickness.
5. Spontaneous Breathing Trail (SBT) Is a process that allows patients to breathe spontaneously with minimal or no ventilatory support for predefined of time (e.g. 30 min) to assess the patient readiness for extubation

ELIGIBILITY:
Inclusion Criteria:

* All mechanically ventilated patients will be:
* Their ages range from 45 to 65 years.
* Their BMI is from 25-29.9kg/m2.
* Mechanically ventilated for at least 24 hours.
* They all have hypoxemic respiratory failure
* Glasgow coma score (GCS) ranged from 6 to 12.
* Richmond Agitation-Sedation Scale score: -2 to +2
* Patients and their relatives had written informed consent.

Exclusion Criteria:

* Hemodynamically unstable patients.
* Patients with rib fractures.
* Patients with implanted pacemaker.
* Obese (BMI greater than 30 kgm2).
* Tachycardia.
* Uncontrolled hypertension.
* History of neuromuscular disease at admission.
* Spinal injuries.
* Inability to trigger mechanical ventilation
* Pregnancy
* An anticipated stay on the ventilator <72 h at the time of study
* Patients who cannot attach electrodes due to local skin damage or infection
* Patients with Severe intestinal gas accumulation, structural abnormalities, and other reasons that prevent ultrasound detection of diaphragm movement.
* Congenital myopathies or neuropathies, and contraindications for expiratory muscle FES (cardiac pacemaker, refractory epilepsy, recent (< 4 weeks) abdominal surgery).
* Patients with unrelieved pneumothorax and restricted diaphragm movement disorders.
* Chest or diaphragm malformation

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
pH (arterial blood gas) | Baseline (within 24 hours prior to intervention) and at successful weaning from mechanical ventilation (within 24 hours of extubation).
PaO₂ (mmHg, arterial blood gas) | Baseline (within 24 hours prior to intervention) and at successful weaning from mechanical ventilation (within 24 hours of extubation).
PaCO₂ (mmHg, arterial blood gas) | Baseline (within 24 hours prior to intervention) and at successful weaning from mechanical ventilation (within 24 hours of extubation).
SaO₂ (%) | Baseline (within 24 hours prior to intervention) and at successful weaning from mechanical ventilation (within 24 hours of extubation)
HCO₃ (mmol/L, arterial blood gas) | Baseline (within 24 hours prior to intervention) and at successful weaning from mechanical ventilation (within 24 hours of extubation)

SECONDARY OUTCOMES:
Diaphragmatic Excursion | Baseline at the start of the study "baseline" and after Successful weaning from mechanical ventilation
Diaphragmatic Fractional Thickness | Baseline at the start of the study "baseline" and after Successful weaning from mechanical ventilation
Abdominal Muscles Wall Thickness | Baseline at the start of the study and after Successful weaning from mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Sherine H Mehani, Professor, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Beni-Suef, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No